CLINICAL TRIAL: NCT06526507
Title: PrEPARE-SCALE: Scaling up Integrated PrEP Delivery in Kenyan Maternal and Child Health Clinics for Pregnant and Postpartum Women
Brief Title: PrEPARE-SCALE: Scaling up Integrated PrEP Delivery in Kenyan Maternal and Child Health Clinics
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anjuli Wagner, Assistant Professor, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00019007; R01MH135730 (NIH)
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Difference in differences design, also known as a controlled pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation strategy package (Experimental): Package includes a Community of Practice, a quality improvement (QI) practice, and a training & delivery toolkit.
  Interventions: Other: Implementation strategy package
- Comparison (No Intervention)

INTERVENTIONS:
Other: Implementation strategy package — Package includes a Community of Practice, a quality improvement (QI) practice, and a training & delivery toolkit.
  Arms: Implementation strategy package

SUMMARY:
This project aims to develop a community of practice; then test a combination of community of practice, quality improvement, and a training toolkit, to enhance implementation and clinical outcomes; and identify patterns attributes associated with successful implementation.

DETAILED DESCRIPTION:
Aim 1: To develop and determine the impact of a Community of Practice (CoP) on stakeholder and healthcare worker engagement and knowledge of integrated pre-exposure prophylaxis (PrEP) delivery.

Aim 2: To determine the impact of a 3-component scale-up package on implementation outcomes and PrEP patient outcomes among pregnant and postpartum populations.

Aim 2a: To determine the impact of the scale-up package on PrEP implementation outcomes, including reach, service penetration, adoption (primary outcomes), and PrEP fidelity and maintenance (secondary outcomes).

Aim 2b: To determine the impact of the scale-up package on PrEP patient outcomes, including PrEP initiation and continuation.

Aim 3: To identify difference-making bundles of facility- and regional-level attributes and implementation processes that influence reach, fidelity implementation, and maintenance.

ELIGIBILITY:
Inclusion Criteria:

Health Care Workers:

* work at a facility involved in study
* involved in PrEP service delivery
* >=18 years

Clients:

* female clients seeking health services at study facilities
* pregnant or postpartum
* >15 years (includes emancipated minors)

Exclusion Criteria:

* N/A

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Service penetration | 1 year
  Number and proportion of pregnant and postpartum maternal child health clinic (MCH) clients who are screened for PrEP
Reach | 1 year
  Number of pregnant and postpartum MCH clients initiated on PrEP each month
Adoption (provider) | 1 year
  Number, proportion, and representativeness of nurses and HIV testing services (HTS) providers who have begun offering or counseling on PrEP in MCH
Adoption (facility) | 1 year
  Proportion of facilities per county that have begun offering PrEP in MCH

CONTACTS AND LOCATIONS:
Overall Officials: Anjuli Wagner, PhD, Principal Investigator — University of Washington
Locations (5):
- Kenya (5):
  - Kapsabet County Referral Hospital, Kapsabet, Nandi
  - Kitale County Referral Hospital, Kitale, Trans Nzoia
  - Uasin Gishu District Hospital, Eldoret, Uasin Gishu County
  - Busia County Referral Hospital, Busia
  - Kenyatta National Hospital, Nairobi